CLINICAL TRIAL: NCT01255150
Title: Frequency of Epidermal Growth Factor Receptor Mutations in Latinos/Hispanics With Non-Small Lung Cancer
Brief Title: Frequency of EGFR Mutations in Latinos/Hispanics With Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110044; 11-C-0044
Record Dates: First submitted 2010-12-04; First posted 2010-12-07 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2015-04-29

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Genetic Ancestry Analysis; Molecular Profiling; Smoking Status; Wood Smoke Exposure; EGFR Mutation Analysis; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Research has shown that the Epidermal Growth Factor Receptor (EGFR) gene is an important target for personalized lung cancer treatment. Individuals who have mutations in the EGFR gene have better responses when treated with certain personalized or targeted therapies compared with conventional chemotherapy. These mutations are more frequent in females with lung cancer who have never smoked, and different ethnic groups have different levels of frequency of the mutations. Researchers are interested in collecting more information on EGFR genetic mutations in Hispanics/Latinos with lung cancer, comparing the frequency of these mutations in males and females and smokers and nonsmokers. This study may lead to better, more personalized care approaches for all individuals with lung cancer.

Objectives:

- To study the frequency of Epidermal Growth Factor Receptor mutations in Hispanic/Latino individuals who have been diagnosed with non-small cell lung cancer.

Eligibility:

- Hispanic or Latino individuals who have been diagnosed with non-small cell lung cancer and who have lung tissue from a previous biopsy or surgery available for research purposes.

Design:

* Participants will provide consent for researchers to examine lung tissue collected from a previous biopsy or surgery.
* Treatment will not be provided as part of this protocol.

DETAILED DESCRIPTION:
Background:

* There is a growing body of evidence that points to genetic heterogeneity of the EGFR pathway in non-small cell lung cancer among different ethnic groups and that underscores the need for consideration of these differences in patient management and in the design of future trials of agents that target the EGFR pathway.
* Activating mutations in EGFR have been found in about 15% of NSCLC patients from North America and Europe, 40% of Asian and 2% in African-Americans.
* However, there is no data on the frequency of EGFR mutations in U.S. Hispanic and Latin American patients with NSCLC.

Primary Protocol Objectives:

* To determine the frequency of EGFR mutations in Hispanic/Latinos with non-small cell lung cancer according to gender and smoking status.
* To study the association between the frequency of EGFR mutations and the percentage of American Indian ancestry, as defined by genetic ancestry analysis, in Hispanic/Latinos with non-small cell lung cancer.

Secondary Protocol Objectives:

-To evaluate the association between EGFR mutations and other clinical variables such as wood smoke exposure, age, stage at presentation, nationality and response to EGFR TKIs.

Eligibility:

* Hispanic or Latino patients with histologically confirmed non-small cell lung cancer.
* Tissue samples from Hispanic or Latino individuals with histologically confirmed non-small cell lung cancer

Design:

* Paraffin embedded tumor samples from Latino patients with non-small cell lung cancer will be collected at the NIH s clinical center and the participating institutions.
* Samples and clinical data will then be sent to the molecular pathology laboratory for EGFR mutation analyses. The remainder DNA will then used for genetic ancestry analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Hispanic or Latino* patients with histologically confirmed non-small cell lung cancer.

Hispanic or Latino* patients with histologically confirmed non-small cell lung cancer.

* For the purpose of this study, the terms Hispanic or Latino is defined as an individual who either self identifies as Hispanic or Latino or was born in any Latin American country.

Tumor samples from deceased Hispanic or Latino individuals with histologically confirmed non-small cell lung cancer for which basic clinical information is available

Pathological waste or surplus stored identified or coded non-small cell lung cancer specimens from Hispanic or Latino individuals for which there is linked clinical information but the location of the person is not feasible to determine.

EXCLUSION CRITERIA:

Patients born in Europe, Asia, Africa or Australia are excluded.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-12-01; Study Completion 2015-04-29

PRIMARY OUTCOMES:
Frequency of EGFR mutations in Hispanic/Latinos with nonsmall cell lung cancer according to gender and smoking status | At tissue and data acquisition upon enrollment
Association between the frequency of EGFR mutations and the percentage of American Indian ancestry, as defined by genetic ancestry analysis, in Hispanic/Latinos with non-small cell lung cancer | At tissue and data acquisition upon enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (12):
- United States (5):
  - Denver Health Medical Center, Denver, Colorado
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Kettering Health Network, Kettering, Ohio
  - Oregon Health and Sciences Universtiy Cancer Center, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Universidad Mayor de San Simon, Cochabamba, Bolivia
- Mexico (4):
  - Universidad de Colima, Colima
  - Instituto Nacional de Cancerologia, Mexico City
  - Center for Research & Development in Health Sciences, Monterrey
  - Universidad Autonoma de Queretaro, Querétaro
- Instituto Nacional de Enfermedades Neoplasicas (INEN), Lima, Peru
- Instituto de Oncologia Luis Razetti, Caracas, Venezuela

REFERENCES:
- [Background] Farjah F, Wood DE, Yanez ND 3rd, Vaughan TL, Symons RG, Krishnadasan B, Flum DR. Racial disparities among patients with lung cancer who were recommended operative therapy. Arch Surg. 2009 Jan;144(1):14-8. doi: 10.1001/archsurg.2008.519. PMID 19153319
- [Background] Wisnivesky JP, McGinn T, Henschke C, Hebert P, Iannuzzi MC, Halm EA. Ethnic disparities in the treatment of stage I non-small cell lung cancer. Am J Respir Crit Care Med. 2005 May 15;171(10):1158-63. doi: 10.1164/rccm.200411-1475OC. Epub 2005 Feb 25. PMID 15735053
- [Background] Clegg LX, Li FP, Hankey BF, Chu K, Edwards BK. Cancer survival among US whites and minorities: a SEER (Surveillance, Epidemiology, and End Results) Program population-based study. Arch Intern Med. 2002 Sep 23;162(17):1985-93. doi: 10.1001/archinte.162.17.1985. PMID 12230422